CLINICAL TRIAL: NCT00652964
Title: PHOX2B Mutation-Confirmed Congenital Central Hypoventilation Syndrome in A Chinese Family: Presentations From Newborn to Adulthood
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200801064R
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Central Alveolar Hypoventilation Syndrome
Keywords: sleep apnea, PHOX2B, hypoventilation, polysomnography
MeSH Terms: conditions — Sleep Apnea, Central; Sleep Apnea Syndromes; Hypoventilation

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation: a family of congenital central hypoventilation syndrome
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — CPAP treatment for patients with congenital central hypoventilation syndrome

SUMMARY:
Detect the PHOX2B Mutation-confirmed congenital central hypoventilation syndrome

DETAILED DESCRIPTION:
Background: Congenital central hypoventilation syndrome (CCHS) is characterized by compromised chemo-reflexes that results in hypoventilation during sleep. Recently, a heterozygous PHOX2B gene mutation was identified in CCHS. This report was made to increase physicians' awareness of this rare disease.

Methods: A Chinese family of CCHS with presentations from newborn to adulthood and genetic analysis confirming the PHOX2B mutation was analyzed. After identifying central hypoventilation in an adult male (index case), clinical evaluation was performed on the complete family, which consisted of the parents, five siblings, and five offsprings. In addition, pulmonary function test, overnight polysomnography, arterial blood gas, and hypercapnia ventilatory response, and genetic screening for PHOX2B gene mutations were performed on living family members.

ELIGIBILITY:
Inclusion Criteria:

* Members of familiar congenital central hypoventilation syndrome

Exclusion Criteria:

* Refuse to participate study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A Chinese family of CCHS with presentations from newborn to adulthood and genetic analysis confirming the PHOX2B mutation was analyzed. After identifying central hypoventilation in an adult male (index case), clinical evaluation was performed on the complete family, which consisted of the parents, five siblings, and five offsprings. In addition, pulmonary function test, overnight polysomnography, arterial blood gas, and hypercapnia ventilatory response, and genetic screening for PHOX2B gene mutations were performed on living family members.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
respiratory failure | cross sectional observation

CONTACTS AND LOCATIONS:
Overall Officials: Peilin Lee, M.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Naitonal Taiwan University Hospital, Taipei, Taiwan